CLINICAL TRIAL: NCT00239239
Title: An Open-label, Single-arm Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Darbepoetin Alfa Administered Three Times Per Week for the Treatment of Anemia in Subjects With Non-myeloid Malignancies Receiving Multicycle Chemotherapy
Brief Title: Fractionated Dosing Study: Study to Evaluate Darbepoetin Alfa for the Treatment of Anemia in Subjects With Non-Myeloid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040232
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Non-Myeloid Malignancies; Anemia; Cancer
Keywords: Non-myeloid malignancy; Chemotherapy-induced anemia; Oncology; Clinical Trials; Pharmacokinetics; Darbepoetin alfa; Aranesp; Amgen
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa

ARMS (1):
- test treatment period (Experimental)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — darbepoetin alfa SC dosing 0.45 mcg/kg 3 times per week through study day 40. Optional extended treatment period: 200 mcg Q2W through study day 110

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics/pharmacodynamics (PK/PD) of darbepoetin alfa administered at a subcutaneous (SC) dose of 0.45 mcg/kg three times weekly (TIW) in anemic patients with non-myeloid malignancies receiving multicycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-myeloid malignancy
* Currently receiving 3-week cyclic chemotherapy treatment with a minimum of 2 additional cycles of chemotherapy planned at the time of enrollment
* Anemia predominately due to cancer or chemotherapy (Hb >= 9.0 and < 11.0 g/dL) at the time of screening
* 18 years of age or older at the time of screening
* Eastern Cooperative Oncology Group (ECOG) score 0-2
* Adequate liver and kidney function Exclusion Criteria:
* Known primary hematologic disorder, which could cause anemia, other than non-myeloid malignancies
* History of chronic myeloid leukemia (CML), acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), acute lymphocytic leukemia (ALL), hairy cell leukemia, Burkitt's lymphoma, or lymphoblastic lymphoma
* Serum folate <= 2.0 ng/mL or vitamin B12 <= 200 pg/mL at screening (anemia related to nutritional deficiencies)
* Iron deficiency [transferrin saturation (TSAT) < 15% and serum ferritin < 10 ng/mL] at screening
* Other diagnoses not related to cancer or chemotherapy, which cause anemia (ie, hemolysis, bleeding, sickle cell anemia)
* Clinically significant inflammatory disease as determined by the investigator (eg, rheumatoid arthritis, Crohn's disease)
* Clinically significant co-morbid medical or psychiatric conditions that may impact subject safety or confound the ability to evaluate study endpoint as determined by the investigator
* Unstable or uncontrolled cardiac disease or condition (ie, angina, congestive heart failure, or cardiac arrhythmia)
* Diastolic blood pressure > 100 mmHg at screening
* Known hypersensitivity of erythropoietic-stimulating proteins (ESPs) or any excipients
* Known history of pure red cell aplasia
* Known positive antibody response to an ESP
* Use of investigational agents not approved or any indication during the previous 30 days prior to enrollment
* ESP therapy (i.e., recombinant human erythropoietin [rHuEPO] or darbepoetin alfa) within 21 days prior to screening or between screening and the first dose of study drug
* RBC transfusion(s) within 21 days prior to screening
* Pregnant or breast-feeding women - Previously enrolled in this study
* Known to be HIV, hepatitis B or C positive
* Any disorder that would compromise the ability of the subject to give written informed consent and comply with study requirements and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-08; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To characterize the PK of darbepoetin alfa administered at a SC dose of 0.45 mcg/kg TIW in the treatment of anemia in subjects with non-myeloid malignancies receiving multicycle chemotherapy | 18 weeks

SECONDARY OUTCOMES:
To assess the effect of darbepoetin alfa treatment on hematopoietic response, red blood cell (RBC) transfusion requirements, and the safety of darbepoetin alfa in subjects receiving multicycle chemotherapy | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com